CLINICAL TRIAL: NCT01525121
Title: Expiratory Rib Cage Compression Does Not Improve Secretion Clearance and Respiratory Mechanics in Mechanically Ventilated Patients
Brief Title: Expiratory Rib Cage Compression in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Fernando Silva Guimaraes, Associate Professor, Centro Universitário Augusto Motta
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MTC_MV
Record Dates: First submitted 2012-01-28; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Pulmonary Infection
Keywords: mechanical ventilation; chest physiotherapy; critical care; pneumonia; Mechanically ventilated patients with pulmonary infection.
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expiratory Rib Cage Compression (Experimental): This a crossover study, so all subjects performed both, control and experimental interventions. The patients were kept in supine at 30 degree head-up position. Ventilatory mode was changed to volume-controlled, with a tidal volume of 8mL/kg, inspiratory flow of 60 Lpm and positive end expiratory pressure (PEEP) of 5 cmH2O. A first tracheal suctioning was done, and the mucus was discarded. Then, a series of two minutes of bilateral expiratory rib-cage compressions ensued. Aiming to minimize inter-therapist variability, the maneuver was applied by the same registered and trained physiotherapist. Control intervention followed the same sequence, but instead of the compressive maneuver they were kept on normal ventilation with the parameters described above.
  Interventions: Other: Expiratory Rib Cage Compression
- Control (No Intervention): This a crossover study, so all subjects performed both, control and experimental interventions. The patients were kept in supine at 30 degree head-up position. Ventilatory mode was changed to volume-controlled, with a tidal volume of 8mL/kg, inspiratory flow of 60 Lpm and positive end expiratory pressure (PEEP) of 5 cmH2O. A first tracheal suctioning was done, and the mucus was discarded. Then, a series of two minutes of bilateral expiratory rib-cage compressions ensued. Aiming to minimize inter-therapist variability, the maneuver was applied by the same registered and trained physiotherapist. Control intervention followed the same sequence, but instead of the compressive maneuver they were kept on normal ventilation with the parameters described above.

INTERVENTIONS:
Other: Expiratory Rib Cage Compression — The therapist hands were positioned on the lower ribs, and the force was applied every two breaths only during the expiration, synchronizing the maneuver rate with the patient's respiratory rate. Then, the patients underwent a suctioning procedure, and a hyperinflation maneuver consisting of a 10 minutes period under pressure support ventilation of 35 cmH2O was done. In control intervention instead of the compressive maneuver the patients were kept on normal ventilation.
  Other Names: Manual thoracic compression
  Arms: Expiratory Rib Cage Compression

SUMMARY:
This is a randomized crossover study, designed to evaluate if the manual expiratory rib cage compression technique improves respiratory mechanics and is effective in secretion removal in mechanically ventilated patients.

DETAILED DESCRIPTION:
Chest physiotherapy is an essential component of the multidisciplinary approach in critical care settings. In this context, a number of devices and manual techniques have been used to remove pulmonary secretions and re-expand collapsed areas. This study was designed to evaluate whether manual rib cage compression improves airway clearance and respiratory mechanics in mechanically ventilated patients. In a randomized crossover trial, 20 mechanically ventilated patients underwent thoracic manual compression and control intervention (normal ventilation) at the same day. The main outcomes were sputum production and the changes in respiratory mechanics.

ELIGIBILITY:
Inclusion Criteria:

* patients under mechanical ventilation
* diagnosis of pulmonary infection
* hypersecretive (defined as the interval between tracheal suctioning < 2 hours)

Exclusion Criteria:

* haemodynamic instability (defined by heart rate > 130 bpm and mean arterial pressure < 60 mmHg)
* use of vasopressor drugs
* absence of respiratory drive
* acute bronchospasm
* acute respiratory distress syndrome
* atelectasis (identified by an independent radiologist that was not participating in the study)
* untreated pneumothorax
* lung haemorrhage.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Sputum Volume (mL) | Day 1

SECONDARY OUTCOMES:
Respiratory Mechanics | Day 1
  Static and effective compliance of the respiratory system Total resistance of the respiratory system

CONTACTS AND LOCATIONS:
Overall Officials: Fernando S Guimarães, PhD, Study Chair — Centro Universitário Augusto Motta; Sara LS Menezes, PhD, Principal Investigator — Centro Universitário Augusto Motta; Agnaldo J Lopes, PhD, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Guimaraes FS, Lopes AJ, Constantino SS, Lima JC, Canuto P, de Menezes SL. Expiratory rib cage Compression in mechanically ventilated subjects: a randomized crossover trial [corrected]. Respir Care. 2014 May;59(5):678-85. doi: 10.4187/respcare.02587. Epub 2013 Oct 8. PMID 24106324